CLINICAL TRIAL: NCT03286205
Title: A Randomized Study to Compare the Dosing Schedule of INFeD in Anemic Patients.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: IP unavailable at site.
Sponsor: Sutter Gould Medical Foundation (Other)
Responsible Party: Principal Investigator, David Adkins, Principal Investigator, Sutter Gould Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Anemia, Iron Deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferryl iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Weekly Dosage (Active Comparator): weekly dose of 100mg
  Interventions: Drug: IV iron
- 3 week dosage (Active Comparator): every 3 week dosage.
  Interventions: Drug: IV iron

INTERVENTIONS:
Drug: IV iron — IV iron infusion based on weekly or every 3 week dosage.

SUMMARY:
The purpose of this study is to establish which dosing schedule of INfed (Iron dextrose) is superior for the treatment of iron deficient anemia.

DETAILED DESCRIPTION:
The purpose of this study is to establish which dosing schedule of INfed (Iron dextrose) is superior for the treatment of iron deficient anemia. The two dosing regimens under review are a low dose weekly or a larger dose given every three weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 18 years old.
2. Being treated by a Sutter Health Physician.
3. Hemoglobin of < 10mg/dl for Men and Women
4. Ferritin </= 10ng/ml
5. Patients in whom oral administration is unsatisfactory or impossible.

Exclusion Criteria:

1. Patients with a history of receiving iron or other hematinic in the preceding 3 months, oral iron is allowable.
2. Anemia due to acute blood loss; menorrhagia is allowed.
3. Patients with a current illness known to interact with iron status.
4. Patients unwilling to consent to required blood draws.
5. Patients who are viewed as unable to complete treatment, based on PI recommendation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
superior dosing regimen exists for INfed | 3 years
  shown by a 2gm/dl increase in HgB
High Dose Effect | 3 years
  INfed can be given at high dose without an increase in AE and/or SAEs frequency

CONTACTS AND LOCATIONS:
Overall Officials: David Adkins, MD, Principal Investigator — Principal Investigator
Locations (1):
- Sutter Gould Medical Foundation, Modesto, California, United States

IPD SHARING:
Plan to Share IPD: No